CLINICAL TRIAL: NCT07161141
Title: Developing an Immersive Virtual Reality Platform to Support Birth Preparedness and Mental Wellbeing in Pregnant Women
Brief Title: Developing an Immersive Virtual Reality Platform
Acronym: VR Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Vesile Koak, Dr, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03072025
Record Dates: First submitted 2025-08-07; First posted 2025-09-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy; Mental Health (Depression); Childbirth Preparation Program
Keywords: Virtual reality; immersive; childbirth; mental health; pregnancy
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): According to international guidelines (e.g., WHO, ACOG, APA), consistent and frequent antenatal care contacts are recommended throughout pregnancy. While a specific number of sessions is not always defined, these guidelines emphasize the importance of providing information within the framework of birth preparedness and complication readiness during these visits. Furthermore, childbirth education programs are encouraged to incorporate psychoeducation and mindfulness-based approaches to support maternal psychological well-being and informed decision-making. In the systematic review, all included studies showed positive effects of the VR and gamification interventions used, regardless of the frequency, intensity, or duration of the intervention (Jingili et al., 2023). VR program will be implemented three times between 20-36 week. Each session will last approximately 10-20 minutes.
  Interventions: Device: Immersive Virtual Reality Platform to Support Birth Preparedness and Mental Wellbeing
- Control (No Intervention): The control group will receive only routine antenatal care, and will complete the pre-test and post-test questionnaires without participating in the intervention.

INTERVENTIONS:
Device: Immersive Virtual Reality Platform to Support Birth Preparedness and Mental Wellbeing — The VR-based intervention will be grounded in a childbirth education framework designed to enhance women's awareness of their attitudes toward childbirth, their readiness for the birthing process, and their expectations related to labor, delivery, and the postpartum period. The program aims to strengthen emotional insight and coping capacities by guiding participants to reflect on their feelings and thoughts throughout the childbirth journey. The intervention will integrate key components such as breath awareness exercises, coping techniques, and motivational messages. While participants receive structured childbirth education, they will simultaneously be supported in developing psychological preparedness through immersive and reflective experiences tailored to foster emotional resilience and self-efficacy.
  The digital labyrinth will be designed both visually and functionally to facilitate immersive navigation. It will be set in an expansive virtual landscape enriched with natural elem
  Arms: Experiment

SUMMARY:
This study is a two-stage, mixed-method, pre-test post-test design aimed at developing and testing an immersive VR intervention for new mothers. This research is 2-arm a 4-week prospective randomized clinical trial

DETAILED DESCRIPTION:
This is an intervention-based study. The first phase of the research will focus on developing the intervention, which will involve the creation of a virtual labyrinth. The concept of "Labyrinth of Birth," was popularized by Pam England. This approach uses the labyrinth as a metaphor to represent the emotional and psychological journey of labor and childbirth. In this model, the mother mentally "walks" through a labyrinth, symbolizing the unique challenges, introspections, and transformations of labor (England, 1998). In this study, the period from pregnancy to birth will be represented as a labyrinth walk with the education, self awarness and motivation content. The content will focus on how to best prepare the mothers during this journey. The content will be revised and finalized based on expert feedback panel, including academics with expertise in pregnancy, childbirth, mental health, VR, until it is deemed appropriate. Then the content will be transferred to a the VR environment. An expert team will be assembled to design the digital labyrinth, and it will be made accessible through VR HMDs. The second phase of the study will focus on testing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The pregnant women between the ages of 18-49
* Primiparous
* At least 20 weeks of gestation
* Single pregnancy
* Without any visual and hearing problems andcan communicate verbally are included to this study.

Exclusion Criteria:

* Pregnant women with multiple pregnancies were multiparous
* Risky pregnancy, and did not accept participation in the study will excluded from the study.
* Individuals with a history of any psychiatric disorder (eg, mood disorder or anxiety disorder) will excluded from this study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 68 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Childbirth Self-Efficacy Scale - Short Form | 4 weeks
  Designed by Lowe in 1993 (Lowe, 1993)to measure the selfconfidence and coping skills of women, CBSEI, consisting of 62 items, was reduced to 32 items by Ip, Chung and Tang in 2008 (Ip et al., 2008). Outcome Expectancy (OE): 16 items evaluating the belief that specific behaviors will lead to desired outcomes during childbirth. The questions in the 10 point Likert type scale are scored between 1 and 10. The scale consists of two subdimensions, each containing 16 questions: "Result Expectation" and "Efficacy Expectation". Self-Efficacy Expectancy (EE): 16 items assessing the confidence in one's ability to perform those behaviors effectively. Scoring: Each item is rated on a 10-point Likert scale, with higher scores indicating greater self-efficacy. The CBSEI scales have excellent internal consistency reliability (.86 to .96)
Childbirth Self-Efficacy Scale - Short Form | From enrollment to the end of the intervention at 4 weeks
  Designed by Lowe in 1993 (Lowe, 1993)to measure the selfconfidence and coping skills of women, CBSEI, consisting of 62 items, was reduced to 32 items by Ip, Chung and Tang in 2008 (Ip et al., 2008). Outcome Expectancy (OE): 16 items evaluating the belief that specific behaviors will lead to desired outcomes during childbirth. The questions in the 10 point Likert type scale are scored between 1 and 10. The scale consists of two subdimensions, each containing 16 questions: "Result Expectation" and "Efficacy Expectation". Self-Efficacy Expectancy (EE): 16 items assessing the confidence in one's ability to perform those behaviors effectively. Scoring: Each item is rated on a 10-point Likert scale, with higher scores indicating greater self-efficacy. The CBSEI scales have excellent internal consistency reliability (.86 to .96)

IPD SHARING:
Plan to Share IPD: No